CLINICAL TRIAL: NCT02089893
Title: Study of the Incidence of Cilioretinal Arteries in the Hungarian Population
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Assistant Professor, Semmelweis University
Other Study IDs: CRA-8504-1/2014/EKU
Record Dates: First submitted 2014-03-15; First posted 2014-03-18 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Cilioretinal Arteries
MeSH Terms: interventions — Fluorescein Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy subjects: Healthy subjects
  Interventions: Device: Fundus photography

INTERVENTIONS:
Device: Fundus photography — Non-mydriatic fundus photographs

SUMMARY:
The purpose of this study is to analyze the retinal arteries, to investigate the incidence, number, types, distribution and localization of cilioretinal arteries in the Hungarian Caucasian population.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian race
* Signed informed consent

Exclusion Criteria:

* Optical media opacities of the eye

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young population
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Incidence of cilioretinal arteries | Through study completion, 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Schneider, MD, PhD, Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University, Department of Ophthalmology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No